CLINICAL TRIAL: NCT03785808
Title: The Impact of Diet Quality on Biomarkers Associated With Lung Cancer Outcomes: Reducing Insulin, Growth Hormones, and Tumors (RIGHT Study)
Brief Title: Reducing Insulin, Growth Hormones, and Tumors
Acronym: RIGHT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to lack of accrual/enrollment
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RG1001909; 8680 (Other: FHCRC)
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Diet Modification; Lung Cancer
Keywords: ketogenic diet; low-fat diet
MeSH Terms: conditions — Lung Neoplasms | interventions — Diet; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be randomized to the low-carbohydrate diet (Diet A), the low-fat diet (Diet B), or the USDA control diet (Diet C). Participants will not be informed about the nature of the intervention diets or the hypotheses we aim to test. The participants will know the diets only as "Diet A", "Diet B", and "Diet C". They will be de-briefed about the nature of the diets and our hypotheses by mail after the study has been completed. At that time, we will also offer them a folder with the dietary guidelines and recipes for the diets they had not been randomized to. The reason participants will be blinded about the diets is that knowing the details may create a placebo effect and/or opting into another intervention diet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diet A (low carbohydrate) (Experimental): Dietary Intervention A will be a low-carbohydrate/high fat, ketogenic-type diet. The diet will include salads, leafy green and non-starchy vegetables, nuts and seeds, eggs, fish and shellfish, and meats in most meals. Grains and added sugars will be excluded, and starchy vegetables, fruits, berries, and legumes will be limited to below 10% of total calorie intake. In addition full fat yogurt, cheeses, and butter will be allowed in moderate amounts. Participants will be encouraged to eat freely from whole-foods rich in fats such as avocados, nuts, seeds, olives, coconut and to use coconut, medium-chain triglyceride (MCT), olive, and avocado oils for cooking and baking on that diet. Participants will aim to fulfill at least 65% of their total calorie requirements from fats.
  Interventions: Behavioral: Special Diet Therapy (low-carb)
- Diet B (low fat) (Experimental): Dietary Intervention B will be low-fat, high carbohydrate whole-foods, plant-based diet. Most animal products and concentrated plant-based protein sources (such as soy isolates) will be excluded. Whole grains, particularly in their cooked form, legumes, vegetables, and fruits will be encouraged while excluding added sugars and refined grains. Added fats and oils will be discouraged on this diet as dietary fat should comprise less than 10% of total energy. Participants can eat freely from all types of fruits, vegetables, and cooked whole grains. Legumes will be emphasized as a replacement for meat and dairy products. Proteins similar to beef, pork, poultry, and dairy products, should be strictly limited, while lean proteins such as eggs, fish, and shellfish may be included occasionally.
  Interventions: Behavioral: Special Diet Therapy (low-fat)
- Diet C (USDA control) (Active Comparator): The control dietary intervention will be based on the 2015 USDA Dietary Guidelines for Americans, with a slightly higher amount of protein than recommended for the general population, and will be comprised of grains (of which ~50% should be consumed as whole grains), 3 servings per day of non-fat or low-fat dairy, legumes, fruit, vegetables, fish, vegetable oils and margarines, and limited quantities of meat, eggs, added sugars, nuts/seeds. Participants will be encouraged to reduce sodium intake to less than 2300 mg (1500 mg for participants over 51 yrs. old) per day, and to consume less than 10% of calories from saturated fat.
  Interventions: Behavioral: Special Diet Therapy (USDA control)

INTERVENTIONS:
Behavioral: Special Diet Therapy (low-carb) — Receive dietary guidelines and recipes and consume a low-carbohydrate diet
  Other Names: DIET; Special Diet Therapy
  Arms: Diet A (low carbohydrate)
Behavioral: Special Diet Therapy (low-fat) — Receive dietary guidelines and recipes and consume a low-fat diet
  Other Names: DIET; Special Diet Therapy
  Arms: Diet B (low fat)
Behavioral: Special Diet Therapy (USDA control) — Receive dietary guidelines and recipes and consume USDA control diet
  Other Names: DIET; Special Diet Therapy
  Arms: Diet C (USDA control)

SUMMARY:
The objective of this project is to compare the effect of two widely implemented cancer diets, differing drastically in macronutrient content, on biomarkers of inflammation, compared to a control diet.

Diet A will be a low-carbohydrate, high-fat ketogenic-type diet with an emphasis on whole foods. By limiting carbohydrate, the diet will have an extremely low glycemic load, thereby minimizing diurnal glucose and insulin excursions.

Diet B will be a low-fat, high-carbohydrate whole foods plant-based diet. It will include only fiber-rich, low-glycemic index sources of carbohydrates and largely eliminate animal protein, which will minimize rapid spikes in blood glucose and insulin and the production of IGF-1. This diet is also hypothesized to improve glucose tolerance and insulin sensitivity, which should further help minimize diurnal glycemic and insulinemic excursions.

Both diets will be compared to a control diet based on the 2015 USDA Dietary Guidelines for Americans (Diet C) in patients suffering from advanced lung cancer as they are completing medical therapy.

The overarching hypothesis motivating this work is that a nutrient dense diet that minimizes known factors involved in tumor growth and progression may improve the effectiveness of therapy. Our specific hypothesis is that participants following either of the experimental diets, A or B, will experience a reduction in biomarkers of insulin resistance and chronic inflammation, both of which are known risk factors for progression in lung cancer, and a greater median time to progression compared to those on the control diet (Diet C).

DETAILED DESCRIPTION:
Little is known about the role of diet in the treatment of lung and other cancers, yet physicians are constantly confronted with the question 'what should I eat' by their patients. Very few randomized controlled dietary interventions have been carried out in this population, hence physicians and dietitians must use their best professional judgement to provide nutrition advice to their patients. Because most believe that nutrition is an important part of the treatment process, patients are eager to implement dietary recommendations and take control of this portion of their medical care. As such, upwards of 64% of patients use the internet to access health information related to cancer treatment with nutrition websites being among the most popular sites visited. However, the dietary advice on the internet aimed at cancer patients is highly discrepant, and even so among cancer treatment centers and research institutions. Within the National Comprehensive Cancer Network (NCCN), of which Fred Hutchinson is a member, only 43% (9 of 21 centers) either provide nutritional information on their website or linked to outside websites. Of those, roughly half recommended a low-fat diet during cancer treatment and the other half recommended a calorie-dense eating plan with the inclusion of high-fat foods. Clearly, this presents a potential pitfall for patients as they, without guidance from their physician or dietitian, may follow dietary advice that is misleading or potentially harmful.

While there is a need for further studies to elucidate the role diet plays during the treatment of cancers in general, lung cancer in particular is understudied in comparison to other types of cancers, and presents a unique opportunity to study the impact of diet during treatment. Primarily, lung cancer patients do not typically suffer from constraints to eating that affect colorectal, esophageal, or head/throat/neck cancer sufferers. Therefore, diet interventions using whole-foods may be fairly well tolerated in this population. A review of nutrition interventions in lung cancer patients carried out through October 2012 indicated that only three controlled studies in 149 patients had been completed, all of which used nutritional supplement products to prevent unintentional weight loss. The authors concluded that nutrition interventions in this population are safe and that more research is needed to determine optimal nutrition recommendations for advanced, inoperable lung cancers

. Through the manipulation of diet, it is possible to selectively target key pathways involved in cancer growth and proliferation. For instance, it is known that cancer cells generate energy through the process of anaerobic glycolysis (the Warburg Effect) which relies primarily on glucose as a fuel source. Evidence from in vitro studies of non-small cell lung cancer (NSCLC) suggests that reducing the glucose availability from the diet might be particularly effective in the treatment of squamous cell carcinomas because the glucose transporter (GLUT-1) expression is markedly elevated in these cancer cells and is associated with enhanced uptake of, and dependence upon, glucose. Case-control studies show that dietary glycemic index is strongly associated with squamous cell carcinoma among NSCLC patients, suggesting that dietary strategies that limit carbohydrate may be effective in 'starving' these predominately glycolytic cells. A diet pattern in which overall energy is not limited, but sources of glucose are selectively reduced, is one mechanism by which cancer progression might be abated. Such low-carbohydrate or - in their most extreme form - ketogenic diets, which provide energy primarily from fat and protein while minimizing carbohydrates, are increasingly shown to be therapeutic for the treatment of glioblastoma and other cancers, as well as neurological diseases, including epilepsy, and cardiovascular disease risk factors.

It is also known that activation of the IGF pathway is critical for tumor cell proliferation, invasiveness, and survival in NSCLC and downregulation of this pathway through dietary manipulation might also be an effective means to suppress cancer growth. The insulin-like growth factor-1 receptor (IGF-1R) is abundantly present on surfaces of tumor cells, and high circulating levels of IGF-1, the ligand for the IGF-1R, are a risk factor for future lung malignancy. As individuals who consume diets high in protein from animal sources have greater levels of circulating IGF-1 compared to those consuming a vegetarian/vegan diet, limiting the intake of animal products may be an intriguing dietary strategy that might influence cancer progression. In our lab, we have shown that insulin sensitivity and glucose tolerance improved after subjects adhered to a diet rich in whole grains, legumes, fruits, and vegetables, that excluded refined sources of energy (added sugar, refined grains, added fats and oils) (Kratz et al. unpublished data). This suggests that such a diet would also reduce the diurnal exposure of tumor cells to both glucose and insulin, which would decrease the availability of fuel and growth hormones for cancer cells. Taken together, both low-carbohydrate/ketogenic diets and low-fat, whole foods plant-based diets could plausibly affect pathways involved in cancer growth or progression by minimizing diurnal exposure to glucose, insulin, and IGF-1.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older) receiving treatment at the Seattle Cancer Care Alliance (SCCA)
* Stage IIIB and IV non-small cell adenocarcinoma or squamous cell carcinoma, or small cell lung cancer with advanced disease receiving therapy with systemic treatment
* Body mass index (BMI) >= 20 kg/m^2
* Body weight within 10% of current weight within the 3 months before starting the study
* Able and willing to attend bi-weekly dietary support sessions at the Seattle Cancer Care Alliance (SCCA) during the initial 12-week intervention period
* Willing and able to follow the dietary regimen
* Willing to maintain usual lifestyle habits (other than diet) throughout the study (e.g., physical activity habits)
* Ability to understand, speak, and write in English
* Ability to provide informed written consent

Exclusion Criteria:

* Neuroendocrine large cell carcinoma or atypical carcinoids with metastatic disease
* Small cell lung cancer receiving curative therapy with radiation
* Use of antidiabetic medications or insulin within the last 6 months
* Presence of grade 2 weight loss, cachexia, and/or severe nausea
* Current participation in therapeutic first line trial
* Alcohol intake > 2 drinks per day
* Major dietary restriction, as determined by the researcher
* Other significant health condition as determined by the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
The impact of diet on IL-6 | 24 weeks
  To compare the impact of consuming the three study diets for 24 weeks on the pro-inflammatory mediator IL-6, which is associated with lung cancer progression.
The impact of diet on hsCRP | 24 weeks
  To compare the impact of consuming the three study diets for 24 weeks on the pro-inflammatory mediator hsCRP, which is associated with lung cancer progression.
The impact of diet on adiponectin | 24 weeks
  To compare the impact of consuming the three study diets for 24 weeks on the pro-inflammatory mediator adiponectin, which is associated with lung cancer progression.
The impact of diet on HOMA-IR | 24 weeks
  To compare the impact of consuming the three study diets for 24 weeks on the homeostasis model assessment insulin resistance (HOMA-IR) index, which is associated with lung cancer progression.
The impact of diet on the Glasgow Prognostic Score for cancer outcomes | 24 weeks
  To compare the impact of consuming the three study diets for 24 weeks on the Glasgow Prognostic Score, which is associated with lung cancer outcomes.
The impact of diet on IGF-1 | 24 weeks
  To compare the impact of consuming the three study diets for 24 weeks on circulating levels of IGF-1, which is associated with lung cancer progression.
The impact of diet on IGFBP-3 | 24 weeks
  To compare the impact of consuming the three study diets for 24 weeks on circulating levels of IGFBP-3, which is associated with lung cancer progression.

SECONDARY OUTCOMES:
Change in body weight | 24 weeks
  To compare the impact of consuming the three study diets for 24 weeks on body weight.
Change in compliance | Baseline up to 52 weeks
  To assess the degree of dietary adherence to the three study diets at 12 weeks and 24 weeks following the initiation of the intervention. Dietary compliance measurement: macronutrient intakes (FFQ) within 10% of total energy intake targets
Response rate | At 12 and 24 weeks
  Will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines.
Progression-free survival | Up to 1 year
  Will be assessed by Kaplan-Meier curves.
Overall survival | Up to 1 year
  Will be assessed by Kaplan-Meier curves.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Kratz, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Seattle Cancer Center Alliance, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT03785808/ICF_000.pdf